CLINICAL TRIAL: NCT02059785
Title: Phase ⅡStudy of Pinocembrin Injection to Treat Ischemic Stroke---Randomized, Double-blind, Placebo-controlled, Multicenter Study
Brief Title: Phase ⅡStudy of Pinocembrin Injection to Treat Ischemic Stroke
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPC-HA1301
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2015-10

CONDITIONS: Ischemic Stroke
Keywords: Pinocembrin for Injection; Placebo; mRS
MeSH Terms: conditions — Ischemic Stroke | interventions — pinocembrin; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pinocembrin for Injection (Experimental): 40mg /60mg in 100ml of a solution of 0.9 percent saline,iv.drip bid,14day
  Interventions: Drug: Pinocembrin for Injection
- placebo (Placebo Comparator): 60mg in 100ml of a solution of 0.9 percent saline,iv.drip bid,14day
  Interventions: Drug: Pinocembrin for Injection

INTERVENTIONS:
Drug: Pinocembrin for Injection
  Other Names: DL0108

SUMMARY:
This research is a Randomized, double-blind, placebo-controlled, multicenter clinical study. Chinese subjects with Ischemic Stroke.

DETAILED DESCRIPTION:
Subjects will randomly enter into one of two groups,the period of treatment is 14 days,follow-up to the 90th days.

ELIGIBILITY:
Inclusion Criteria:

* 35-75 hospitalized patients
* Patients with acute stroke ≤24h
* NIHSS score 6-20 at time of enrollment , the score ≥2 of item 5 and/or 6
* For the first time or always without obvious sequelae of stroke disease(mRS≤1）
* Informed consent

Exclusion Criteria:

* The disease such as Acute intracerebral hemorrhage,tumor and encephalitis which cause similar symptoms
* Patient with NIHSS level of consciousness score≥2 or dementia,or other patients who the investigator think that don't fit into the study
* TIA
* Symptoms of disease rapidly improving during the randomized
* Severe hypertension(SBP > 200 mmHg or DBP >110 mmHg)
* Inadequate liver function(AST or ALT greater than 2 times the upper limit of normal values);Renal impairment (Creatinine clearance <60ml/min）
* Severe system or viscera organic disease
* Have used other neuroprotectant or other experimental drugs
* Patient who are unlikely to complete the study that due to a severe clinical condition
* Pregnant or breast-feeding
* Participation in a previous clinical study within 30 days
* Meets all other exclusion criteria

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To determination the proportion of subjects that 0-1 score of mRS after treatment 90 days | 90 days

SECONDARY OUTCOMES:
To compare treatment arms in terms of change from baseline to endpoint in NIHSS score. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yong Jun, Ph.D, Study Director — Beijing Tiantan Hospital affilliated to Capital Medical University
Locations (1):
- Beijing Tiantan Hospital affilliated to Capital Medical University, Beijing, Beijing Municipality, China